CLINICAL TRIAL: NCT04245969
Title: Efficacy of 448kilohertz Capacitive Resistive Monopolar Radiofrequency Stimulation in Chronic Shoulder Pain: A Randomised Controlled Trial
Brief Title: Efficacy of 448kilohertz Capacitive Resistive Monopolar Radiofrequency Stimulation in Chronic Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, SANTIAGO NAVARRO LEDESMA, UNIVERSITY PROFESSOR, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRMRFSP
Record Dates: First submitted 2019-10-15; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Chronic Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- INTERVENTION (Experimental): 448 kilohertz Capacitive Resistive Monopolar Radiofrequency stimulus on the shoulder
  Interventions: Device: Experimental: 448 kilohertz Capacitive Resistive Monopolar Radiofrequency stimulus
- Placebo Monopolar Radiofrequency stimulus (Experimental): To simulate the application of Monopolar Radiofrequency stimulus on the affected shoulder
  Interventions: Other: Sham comparator
- No intervention group (Experimental): To evaluate at the same time than the others groups but without being treated with 448 kilohertz Capacitive Resistive Monopolar Radiofrequency.
  Interventions: Other: No intervention

INTERVENTIONS:
Device: Experimental: 448 kilohertz Capacitive Resistive Monopolar Radiofrequency stimulus — 448kilohertz capacitive resistive monopolar radiofrequency will be applied on the shoulder and thoracic area
  Arms: INTERVENTION
Other: Sham comparator — A simulation of 448kilohertz capacitive resistive monopolar radiofrequency will be carried out to make believe the patient to be treated through this equipment.
  Arms: Placebo Monopolar Radiofrequency stimulus
Other: No intervention — These participants will be assessed at the same time than the rest of participants. They will not receive any kind of treatment.
  Arms: No intervention group

SUMMARY:
448kilohertz capacitive resistive monopolar radiofrequency is a novel technique in physiotherapy and its usefulness and clinical relevance is still to be investigated. Current studies show promising results in different musculoskeletal disorders, however further studies with proper designs and conclusive findings are necessary.

DETAILED DESCRIPTION:
Shoulder pain is is one of the most common musculoskeletal disorders, presenting a high prevalence in primary care centers. Many factors have been proposed as the cause of pain, however it is still controversial and the same regarding the best treatment option.

Treatments throw different techniques have been investigated, showing a variety of results in terms of pain and sensitivity. However, the use of 448kilohertz capacitive resistive monopolar radiofrequency as the focus of the treatment is to be explored.

The hypothesis of the present project is that focus treatments on 448kilohertz capacitive resistive monopolar radiofrequency on the shoulder will produce better outcomes in terms of ultrasound assessment, strength, pain, sensitivity and range of movement, when compared to traditional methods used like manual therapy and/or exercise.

The stimulus will be carried out on the shoulder region (suprascapular, axillar, subscapular, long thoracic or pectoralis nerves) and the thoracic region. All interventions will be developed by the same examiner, who is a physiotherapist with 6 years of clinical experience.

The outcome measures will be electromyography and dynamometry to measure strength and muscular activity. The movements required to the patient will be shoulder flexion, abduction, adduction, and extension.

To quantify sensitivity, pain pressure thresholds will be measured throw an algometer placed on the coracoid process, on the lateral area of the shoulder (two centimeters below the acromion and on the acromioclavicular joint).

To measure the range of movement, a goniometer will be used for both glenohumeral and scapular rotations.

To measure quality of life and psychological factors several questionnaires will be asked (Pain catastrophizing scale, Pain vigilance and awareness questionnaire, Self-efficacy, SPADI, Tampa Scale-11, McGill)

ELIGIBILITY:
Inclusion Criteria:

* To suffer from shoulder pain more than three months.
* Men or women aged between 18 to 65 years;
* Unilateral pain located in the anterior and/or lateral shoulder region;
* 2 out of 3 positive clinical tests (Hawkins-Kennedy; Jobe; Neer);
* Pain with normal activity ≥ 4/10 on a visual analogue scale;
* Nontraumatic onset of shoulder pain.

Exclusion Criteria:

* History of significant shoulder trauma, such as fracture or ultrasonography-clinically suspected full thickness cuff tear, following the classification of Wiener and Seitz
* Recent shoulder dislocation in the past two years
* Systemic illnesses such as rheumatoid arthritis
* Adhesive capsulitis of the shoulder
* Shoulder pain originating from the neck or if there was a neurological impairment, osteoporosis, hemophilia and/or malignancies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-30 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline ultrasound imaging at 3 months | time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)
  Elastography
Change from Baseline ultrasound imaging at 3 months | time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)
  Tendon thickness

SECONDARY OUTCOMES:
Electromyography | time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)
  Electromyography of different shoulder muscles (deltoid, trapezius,serratus )will be measured.
Change from Baseline dynamometry at 3 months | time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)
  Strength of different shoulder muscles (deltoid, trapezius,serratus )will be measured.
Algometry | time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)
  Pain pressure thresholds of different shoulder muscles (deltoid, trapezius,serratus )will be measured
Range of movement | time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)
  Measurement of mobility in different planes:
  Active shoulder flexion and abduction will be measured with the patient seated, in the scapular plane and relative to the thorax. In addition, active external and internal rotation will be measured in neutral (shoulder in adduction), 30°, 60° and 90° of abducted position.
Change from baseline SPADI (Shoulder Pain And Disability Index) questionnaire at three months | time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities.
Catastrophizing Scale questionnaire | time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)
  Assessment of the mechanisms by which catastrophizing impacts on pain experience.
Heart rate variability (HRV) | time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)
  Measurement of Autonomic nervous system activity:
  Resting HRV provides quantitative information regarding cardiac autonomic tone.
Autonomic Symptom Profile questionnaire (ASP) | time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later)
  Measurement of Autonomic nervous system activity:
  The Autonomic Symptom Profile (ASP) is a validated self-report questionnaire that comprehensively assesses autonomic symptoms across 11 subscales and yields a composite autonomic symptom score

IPD SHARING:
Plan to Share IPD: No